CLINICAL TRIAL: NCT00006405
Title: APEX: Adiposity Prevention by Exercise in Black Girls
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 930
Record Dates: First submitted 2000-10-12; First posted 2000-10-13 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
To determine whether a one year afternoon exercise program will reduce adiposity in African American girls, ages 8 to 10.

DETAILED DESCRIPTION:
BACKGROUND:

Obese children who engage in vigorous exercise programs show beneficial effects on total body percent fat (percent BF) and visceral adipose tissue (VAT); however, little is known about how to prevent accretion of total body or visceral adiposity in high risk youths, such as African-American (AA) females.The project has important health implications for two reasons, as follows. There is a dearth of information concerning the effects of exercise interventions in school and community settings. If the study shows that an afternoon exercise program reduces accretion of general and visceral adiposity and has a favorable impact on fitness and health in a population that is at high risk of obesity, then schools may be encouraged to implement similar interventions to prevent juvenile obesity and associated health problems.

The study was awarded in response to a Program Announcement on Physical Activity and Cardiopulmonary Health released in October 1994 jointly by the NHLBI, the National Institute of Diabetes and Digestive and Kidney Diseases, and the National Institute of Nursing Research.

DESIGN NARRATIVE:

The design involves randomization of 200 African American girls, eight to 10 years of age into intervention or control groups. After one year, the groups are compared to test the primary hypothesis that a one year afternoon exercise program will reduce accretion of general and visceral adiposity in these girls. Then the girls will switch group assignments for the next year. The pattern of data over the three time points will show what happens over a two year period in which the youths are, or are not, involved in the exercise program. The measurements will include: (1) percent body fat with dual-energy x-ray absorptiometry; (2) visceral adipose tissue (VAT) with magnetic resonance imaging; (3) cardiovascular fitness with a multi-stage treadmill test; (4) cardiovascular disease (CVD) risk factors (i.e., the ratio of total to high density lipoprotein cholesterol, insulin, systolic blood pressure, and fibrinogen); (5) free-living exercise and diet; (6) psychosocial variables (i.e., self-efficacy and self-concept); (7) sexual maturation; (8) anthropometric measures. The exercise program will be implemented in neighborhood schools for 90 minutes each weekday afternoon. Transportation will be provided if needed. Sessions will include motor skill instruction and aerobic exercises.

ELIGIBILITY:
No eligibility criteria

Ages: 8 Years to 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2002-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paule Barbeau — Augusta University

REFERENCES:
- [Background] Gutin B, Yin Z, Humphries MC, Hoffman WH, Gower B, Barbeau P. Relations of fatness and fitness to fasting insulin in black and white adolescents. J Pediatr. 2004 Dec;145(6):737-43. doi: 10.1016/j.jpeds.2004.07.016. PMID 15580193
- [Background] Gutin B, Yin Z, Humphries MC, Bassali R, Le NA, Daniels S, Barbeau P. Relations of body fatness and cardiovascular fitness to lipid profile in black and white adolescents. Pediatr Res. 2005 Jul;58(1):78-82. doi: 10.1203/01.PDR.0000163386.32348.90. Epub 2005 May 5. PMID 15879296